CLINICAL TRIAL: NCT03593252
Title: Pre-Operative Mechanical Bowel Preparation And Prophylactic Oral Antibiotics For Pediatric Patients Undergoing Elective Colorectal Surgery: A Feasibility Randomized Controlled Trial
Brief Title: Bowel Preparation in Elective Pediatric Colorectal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Collaborators: McMaster Pediatric Surgery Rresearch Collaborative (MPSRC) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Bowel_prep_pediatric_sx
Record Dates: First submitted 2018-05-22; First posted 2018-07-20 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Colostomy; Hirschsprung Disease - Pull Through; Necrotizing Enterocolitis; Inflammatory Bowel Diseases; Meconium Ileus; Bowel Obstruction; Elective Surgery
MeSH Terms: conditions — Enterocolitis, Necrotizing; Inflammatory Bowel Diseases; Meconium Ileus; Intestinal Obstruction | interventions — Sennosides; picosulfate sodium; Magnesium Oxide; Citric Acid; Pico-Salax; Metronidazole; Neomycin; Cefazolin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to the following study arms:
  1. Combination bowel prep: Mechanical preparation and oral non-absorbable antibiotics + standard care.
  2. Oral antibiotics + standard care.
  3. No preparation, with standard care. *Standard care (all groups):
     * Nil per os (NPO) prior to general anesthesia
       * Solids until 8 hours prior to surgery, formula until 6 hours, breast milk until 4 hours, clear fluids until 2 hours
     * Prophylactic IV antibiotics
       * Cefazolin (30mg/kg) and metronidazole (15mg/kg) within 60 minutes of incision
       * Re-dosing if procedure exceeds 4 hours
       * In case of beta-lactam allergy allergy, clindamycin 5mg/kg and gentamicin 7mg/kg will be used.
Who Masked: Outcomes Assessor
Masking Description: The patient's records will mention he/she is part of a study and will mention the study number, while the actual medications received (group allocation) will not be mentioned. The outcome detector, assessing the patient from day 1 in the hospital to the end of the study, will not have access to information on the study group allocation. The statistician analyzing the data will have a coded and de-identified version, and will be blinded to study groups to ensure unbiased analysis.
  For the purpose of blinding the data analyst, data on bowel prep diary will be withheld until analysis for all other outcomes is done and finalized.
  The principle investigators and the research coordinator will be involved in prescribing the prep regimen preoperatively and will not be blinded. The patient and family will be aware of the medications used and will not be blinded either. Also, the pharmacist will have access to the treatment allocation list, and cannot be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Combination bowel prep (Experimental): Patients will received mechanical bowel preparation (age appropriate dose, starting 2 days before surgery) and prophylactic oral antibiotics (3 doses, 1 day before surgery).
  Clear fluids (or breast milk if applicable) will be given starting day before surgery.
  The standard care will also be delivered (NPO for anesthesia and intravenous antibiotics on induction) Patients/parents will be provided with stool diary to document the adequacy of preparation. This will include frequency and character of stool according to Bristol grade. The treating surgeon will rate the adequacy of the preparation intra-operatively.
  Interventions: Drug: Senna; Drug: Sodium Picosulfate, Magnesium Oxide and Citric Acid; Drug: Metronidazole Oral; Drug: Neomycin; Drug: Cefazolin; Drug: Metronidazole; Other: Nil per os; Other: Clear fluids the day before surgery
- Oral antibiotics (Active Comparator): The patients will receive prophylactic oral antibiotics (3 doses, 1 day before surgery)as well as standard care (NPO for anesthesia and intravenous antibiotics on induction).
  Interventions: Drug: Metronidazole Oral; Drug: Neomycin; Drug: Cefazolin; Drug: Metronidazole; Other: Nil per os
- No prep (Placebo Comparator): Patients will receive no pre-operative bowel prep. The will receive the standard care only.
  Interventions: Drug: Cefazolin; Drug: Metronidazole; Other: Nil per os

INTERVENTIONS:
Drug: Senna — Laxative,used for bowel preparation
  Other Names: Senokot
  Arms: Combination bowel prep
Drug: Sodium Picosulfate, Magnesium Oxide and Citric Acid — Laxative used for bowel preparation
  Other Names: Pico-Salax
  Arms: Combination bowel prep
Drug: Metronidazole Oral — Oral antibiotic
  Other Names: flagyl
  Arms: Combination bowel prep; Oral antibiotics
Drug: Neomycin — Oral non-absorbable antibiotic
  Arms: Combination bowel prep; Oral antibiotics
Drug: Cefazolin — Intravenous antibiotic to be given on anesthesia induction and prior to incision as a prophylactic antibiotic.
  Other Names: ancef
Drug: Metronidazole — Intravenous antibiotic to be given on anesthesia induction and prior to incision as prophylactic antibiotic.
  Other Names: Flagyl
Other: Nil per os — Fasting orders according to anesthesia prior to surgery: No solid for >=8 hours, no formula milk/full liquids >= 4hours; no breast milk or clear fluids >=2hours.
  Other Names: NPO
Other: Clear fluids the day before surgery — As part of bowel preparation, participants will be asked to stick to clear fluids following breakfast the day before surgery. Breast milk is allowed if applicable.
  Arms: Combination bowel prep

SUMMARY:
Infections after elective intestinal surgery remain a significant burden for patients and for the health care system. The cost of treating a single surgical site infection is estimated at approximately $27,000. In adult patients, there is good evidence that the combination of oral antibiotics and mechanical bowel preparation is effective at reducing infections after intestinal surgery. In children, the body of evidence is much weaker. In this population, little evidence exists for oral antibiotics reducing infections and no data exists as to the effect of combining antibiotics with mechanical bowel preparation (such as polyethylene glycol (PEG)). The goal of the proposed study is to examine the effects of oral antibiotics with and without the combined use of mechanical bowel preparation on the rate of post-operative infectious complications in children aged 6 months to 18 years. This will be compared to the institution's current standard of care, which is to abstain from any type of mechanical bowel preparations or oral antibiotic administration before intestinal surgery.

DETAILED DESCRIPTION:
Background:

A Cochrane review of randomized controlled trials of MBP use in adults showed no difference in the rate of wound infection or anastomotic leak in colon or rectal procedures with MBP compared to no preparation (Guenaga, Matos, & Wille-Jorgensen, 2011). Two recent systematic reviews and meta-analyses support those findings. Lok and colleagues (2018) identified two randomized controlled trials and four retrospective reviews for patient <21 years, looking at preoperative MBP and its effect on the incidence postoperative complications, including anastomotic leak, wound infection, and intra-abdominal infection (Janssen Lok M 2018). Overall, MBP before colorectal surgery did not significantly decrease the incidence of post-operative outcomes. This was consistent with findings from a systematic review in mechanical bowel preparation in pediatric population. The review showed that the risk of developing a post-operative infection was 10.1% in patients who received MBP compared to 9.1% in patients who did not receive MBP, resulting in no statistically significant difference difference (risk difference of -0.03% (95% CI, -0.09% - 0.03%)) (Zwart 2018).

With regards to OA alone, the adult literature showed promising results in favour of the OA. In a Cochrane review on antimicrobial prophylaxis in colorectal surgery, the addition of OA to the intravenous antibiotics was found to reduce surgical wound infection (RR 0.56, 95% CI 0.43 to 0.74) (Nelson, Gladman, & Barbateskovic, 2014).

There are fewer studies in the pediatric population on the subject, they contain fewer patients and are mainly retrospective in nature. In a multi-center retrospective study, Serrurier et al. (2012), reviewed outcomes in children who underwent colostomy closure, and found higher rates of wound infection (14% vs. 6%, p=0.04) and a longer hospital length of stay in children who received MBP. In a retrospective cohort study including 1581 pediatric patients from PHIS database, post-operative complications were found to be highest in the no preparation group compared to combination prep and OA alone (23.3%, 15.9%, and 14.2% respectively; p=0.002) (Ares 2018). One study compared MBP alone versus MBP with OA in children undergoing colostomy closure post anorectal malformation repair and found no difference in overall SSI rates (MBP+OA: 13% (7/53) versus MBP alone: 17% (7/12) p=0.64) (Breckler, Rescorla, & Billmire, 2010). The authors found that the use of MBP alone was associated with a greater risk of wound infection (14% vs. 6%, p=0.04) and a longer hospital stay. Evidence to support the sole use of oral antibiotics versus in combination with MBP is lacking, particularly in the pediatric literature, with more studies being required to address this question.

One recent meta-analysis including adults assessed 8458 adult patients (38 clinical trials), comparing 4 groups of different bowel preparation: MBP with OA, OA only, MBP only, and no preparation. The primary outcome was the total rate of incisional and organ/space SSIs. Results showed that only MBP with OA versus MBP alone was associated with a statistically significant reduction in SSI rates. The use of OA without MBP was not associated with a statistically significant reduction in SSI rates when compared to any other group. The authors concluded that MBP with OA was associated with the lowest risk of SSI, followed by OA only (Toh et al., 2018).

It remains unclear whether the addition of MBP to OA in pediatric population affects the rate of post-operative infectious complications positively or negatively. The current study is therefore needed to build on the work conducted in the adult literature to determine best practices for the pediatric population.

Purpose:

This is a pilot study to check the feasibility of conducting a randomized controlled trial to assess the efficacy of oral nonabsorbable antibiotics, with or without mechanical bowel preparation, in reducing the rate of post-operative infectious complications occurring within 30 days post-operatively in children and adolescents (aged 6 months to 18 years) undergoing elective colon or rectal surgery.

Post-operative complications include: surgical site infections (incisional, organ-space, and anatomic leak), length of hospital stay, readmission, post-operative use of therapeutic antibiotics, re-operation, occurrence of electrolyte disturbances (in case MBP was used), and occurrence of C. difficile infection.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients aged three months to eighteen years being treated by the Pediatric General Surgery service at McMaster Children's Hospital.
2. Undergoing elective colorectal surgery.
3. Parents or legal guardian able to give free and informed consent.

Exclusion Criteria:

1. Non-elective surgery
2. Procedures that would not require mechanical bowel preparation:

   1. Colorectal resection with an existing diverting small bowel ostomy.
   2. Completion proctectomy - Ileal Pouch Anal Anasotmosis (IPAA)
   3. Closure of small bowel ostomy (e.g. ileostomy)
3. Mechanical bowel obstruction
4. Known hypersensitivity to laxatives or oral antibiotics (neomycin and metronidazole)
5. Contraindication to oral antibiotics
6. Patients on long-term antibiotics for other reasons
7. Congestive heart failure
8. Renal insufficiency
9. Other medical conditions precluding the use of either oral antibiotics or mechanical bowel preparation
10. Co-enrolment in another intervention trial

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility (no. enrolled) | From randomization to 30 days post-operatively
  recruitment rate (percentage of eligible patients enrolled and retained to the end of study).
rate of post-randomization exclusions | From randomization to 30 days post-operatively
  Patients excluded after being randomized
Protocol deviations | From randomization to 30 days post-operatively
  Number of protocol deviations
Adverse events | From randomization to 30 days post-operatively
  Any expected and unexpected adverse event, with grade of adverse event
Incomplete follow-up | From randomization to 30 days post-operatively
  Number missing follow-up appointments at 2 week mark

SECONDARY OUTCOMES:
Superficial Incisional surgical site infection (SSI) | 30 days post-operatively.
  Rate of SI-SSI (superficial or deep, number of patients who developed SSI per group/subgroup).
Deep incisional surgical site infection (SSI) | 30 days post-operatively.
  Rate of DI-SSI (number of patients who developed SSI per group/subgroup).
Organ space - Surgical site infection (SSI) | 30 days post-operatively.
  Rate of OS- SSI (number of patients who developed OS-SSI per group/subgroup).
Anastomotic leak - Surgical site infection (SSI) | 30 days post-operatively.
  Rate of anastomotic leak (verified by a contrast study or intra-operatively) (number of patients who developed OS-SSI per group/subgroup).
Length of hospital stay | 30 days post-operatively.
  Post-operative hospitalization on primary admission in days
Time to full enteric feed. | 30 days post-operatively.
  Post-operative return to full feed/diet in days
Re-admission | 30 days post-operatively.
  admission in post-operative period for a reason related to the surgery (yes/No)
Re-operation | 30 days post-operatively.
  Yes/No. Note:operation indication is directly related to the surgery
Electrolyte disturbance | On day of surgery
  significant changes in electrolytes (abnormal levels) (Yes/No)
Electrolyte disturbance | On day of surgery
  If abnormal levels were detected, whether this was associate by clinical signs (Yes/No)
Clostridium difficile infection | 30 days post-operatively.
  Occurrence of C. difficile infection post-operatively (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa VanHouwelingen, MD, MPH, FRCSC, Principal Investigator — McMaster Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breckler FD, Rescorla FJ, Billmire DF. Wound infection after colostomy closure for imperforate anus in children: utility of preoperative oral antibiotics. J Pediatr Surg. 2010 Jul;45(7):1509-13. doi: 10.1016/j.jpedsurg.2009.10.054. PMID 20638534
- [Background] Guenaga KF, Matos D, Wille-Jorgensen P. Mechanical bowel preparation for elective colorectal surgery. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD001544. doi: 10.1002/14651858.CD001544.pub4. PMID 21901677
- [Background] Julious, S. A. (2005). Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics, 4, 287-291.
- [Background] Nelson RL, Gladman E, Barbateskovic M. Antimicrobial prophylaxis for colorectal surgery. Cochrane Database Syst Rev. 2014 May 9;2014(5):CD001181. doi: 10.1002/14651858.CD001181.pub4. PMID 24817514
- [Background] Rangel SJ, Islam S, St Peter SD, Goldin AB, Abdullah F, Downard CD, Saito JM, Blakely ML, Puligandla PS, Dasgupta R, Austin M, Chen LE, Renaud E, Arca MJ, Calkins CM. Prevention of infectious complications after elective colorectal surgery in children: an American Pediatric Surgical Association Outcomes and Clinical Trials Committee comprehensive review. J Pediatr Surg. 2015 Jan;50(1):192-200. doi: 10.1016/j.jpedsurg.2014.11.028. Epub 2014 Nov 12. PMID 25598122
- [Background] Serrurier K, Liu J, Breckler F, Khozeimeh N, Billmire D, Gingalewski C, Gollin G. A multicenter evaluation of the role of mechanical bowel preparation in pediatric colostomy takedown. J Pediatr Surg. 2012 Jan;47(1):190-3. doi: 10.1016/j.jpedsurg.2011.10.044. PMID 22244415
- [Background] Smith RL, Bohl JK, McElearney ST, Friel CM, Barclay MM, Sawyer RG, Foley EF. Wound infection after elective colorectal resection. Ann Surg. 2004 May;239(5):599-605; discussion 605-7. doi: 10.1097/01.sla.0000124292.21605.99. PMID 15082963
- [Background] Koullouros M, Khan N, Aly EH. The role of oral antibiotics prophylaxis in prevention of surgical site infection in colorectal surgery. Int J Colorectal Dis. 2017 Jan;32(1):1-18. doi: 10.1007/s00384-016-2662-y. Epub 2016 Oct 24. PMID 27778060
- [Background] Janssen Lok M, Miyake H, O'Connell JS, Seo S, Pierro A. The value of mechanical bowel preparation prior to pediatric colorectal surgery: a systematic review and meta-analysis. Pediatr Surg Int. 2018 Dec;34(12):1305-1320. doi: 10.1007/s00383-018-4345-y. Epub 2018 Oct 20. PMID 30343324
- [Background] Zwart K, Van Ginkel DJ, Hulsker CCC, Witvliet MJ, Van Herwaarden-Lindeboom MYA. Does Mechanical Bowel Preparation Reduce the Risk of Developing Infectious Complications in Pediatric Colorectal Surgery? A Systematic Review and Meta-Analysis. J Pediatr. 2018 Dec;203:288-293.e1. doi: 10.1016/j.jpeds.2018.07.057. Epub 2018 Sep 12. PMID 30219553
- [Background] Ares GJ, Helenowski I, Hunter CJ, Madonna M, Reynolds M, Lautz T. Effect of preadmission bowel preparation on outcomes of elective colorectal procedures in young children. J Pediatr Surg. 2018 Apr;53(4):704-707. doi: 10.1016/j.jpedsurg.2017.03.060. Epub 2017 Mar 30. PMID 28433362
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Toh JWT, Phan K, Hitos K, Pathma-Nathan N, El-Khoury T, Richardson AJ, Morgan G, Engel A, Ctercteko G. Association of Mechanical Bowel Preparation and Oral Antibiotics Before Elective Colorectal Surgery With Surgical Site Infection: A Network Meta-analysis. JAMA Netw Open. 2018 Oct 5;1(6):e183226. doi: 10.1001/jamanetworkopen.2018.3226. PMID 30646234
- [Background] Nelson RM, Ross LF. In defense of a single standard of research risk for all children. J Pediatr. 2005 Nov;147(5):565-6. doi: 10.1016/j.jpeds.2005.08.051. No abstract available. PMID 16291339
- [Derived] Briatico D, Flageole H, Al-Shahwani N, Farrokhyar F, VanHouwelingen L. Pre-operative mechanical bowel preparation and prophylactic oral antibiotics for pediatric patients undergoing elective colorectal surgery: a protocol for a randomized controlled feasibility trial. Pilot Feasibility Stud. 2024 May 25;10(1):85. doi: 10.1186/s40814-024-01476-6. PMID 38796500